CLINICAL TRIAL: NCT03678194
Title: Treating Depression on a Day-to-day Basis: Development of a Novel Clinical Tool for Physicians Based on a Smartphone Application, the SMART Project (Smartphones and Mood Disorders, an Application for Research and Treatment)
Brief Title: Treating Depression on a Day-to-day Basis: Development of a Tool for Physicians Based on a Smartphone Application
Acronym: SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018 A01465-50
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Depression; Psychiatric Disorder; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases
Keywords: Depression; Smartphone; Relapse prevention; Mobile support system; eHealth; Ecological; Randomized; Multicentric
MeSH Terms: conditions — Depression; Mental Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: 200 patients with a DSM-V diagnosis of depression are recruited. Patients are randomly assigned to receive either a 6 weeks smartphone application with daily evaluations, or no application.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone application (Experimental): This group of subjects receives mobile support system and conventional treatment (clinical evaluation and follow-up). The smartphone application will be downloaded on patients' smartphone to daily evaluate symptomatology, medication adherence…
  Interventions: Device: Smartphone Support System
- Standard services (No Intervention): This group of patients receives conventional treatment only. Clinical evaluations are provided at the same endpoint. Patients still receive standard services for depression.

INTERVENTIONS:
Device: Smartphone Support System — 6 weeks smartphone application with daily evaluations
  Arms: Smartphone application

SUMMARY:
Testing and validating an e-health (smartphone application) approach to better understand the determinants of day-to-day symptomatology in depression, medication adherence, and treatment efficacy in the goal of maximizing patient care.

DETAILED DESCRIPTION:
In industrialized countries, depression is the leading cause of disability with a cumulative DALY (disability adjusted life years) that his greater than all the other psychiatric or medical conditions (WHO, 2004). Although the medical treatment is efficient for a large number of patients, two major pitfalls can be highlighted: i). the difficulty to identify and alter risk factors related to therapeutic observance; and ii). the heterogeneous presentation of depression, which may require specific interventions depending on the clinical presentation of the patient.

Ecological Momentary Assessment (EMA; also referred to as the Experience Sampling Method) is a method used to gather and interpret real-time data collected in the contexts of daily life through mobile technologies (Stone 1994). It has been used extensively in the field of psychiatry and specifically in mood disorders and it has been shown to be both feasible for patients with depression (Husky 2010, Swendsen 2012) and effective in identifying determinants of mood fluctuations and medication observance (Myin Germeys 2003, Ebner-Primer 2009, Solhan 2009, Silk 2011, Wichers 2010, Rot 2012, Armey 2015, Wenze 2010, Armey 2015). The restitution of the data to patients also has an important added benefit in terms of prognosis, as patients are better integrated in their own care (Wichers 2011, Kramer 2014).

Although EMA has been shown to offer promising advantages, it has also been limited by the technical solutions used to gather information on daily life experiences. Rather than using research-dedicated devices which represent the majority of existing tools, the development of an application-based solution could revolutionize the field by creating the first effective and widely-diffusable tool to help clinicians better manage depression with the collaboration of their patients. This application would be designed to help patients monitor their symptoms, while providing regular interventions to increase medication.

This is a randomized study in two groups to test and validate an e-health (smartphone application) approach to better understand the determinants of day-to-day symptomatology in depression, medication adherence, and treatment efficacy in the goal of maximizing patient care.

In this multicentric study, 200 patients with a DSM-V diagnosis of depression are recruited.

Participants will be assessed by:

* Hetero-evaluations: diagnostic (MINI), depressive symptomatology (HDRS), clinical impression (CGI).
* Auto-evaluations: depressive symptomatology (BDI), medication adherence (MARS), Quality of Life (Q-LES-Q-SF), therapeutic alliance (4PAS).

Two groups will be formed by randomization (100 per groups):

* Groupe SMART: smartphone (experimental group). This group will performed all clinical evaluations and will download the study application on their smartphone to answer daily questionnaires about symptom severity, medication adherence, during 6 weeks. Participants will be given a smartphone, if the subject does not have one. Clinical visits with psychiatrist will be performed every two weeks, with questionnaires to fill.
* Groupe TAU: Treatment as Usual (control group). This group will performed all clinical evaluations and have the same follow-up as the intervention group, but without smartphone application.

Expected results Patient benefit: The principle expected benefit for patients concerns their more active participation in their own health care, in the philosophy that the better they understand their disorder and the triggers of symptom expression, the better than can intervene to improve their mental health.

Clinician benefit: It can provide high resolution data of depressive symptoms, therapeutic adherence and symptoms fluctuations on his patients, to better follow the remission or to adjust treatment daily dose.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years;
* Fulfilling the Diagnostic and Statistical Manual version IV (DSM-IV) criteria of depression assessed by the Structured Clinical Interview;
* Patients started their antidepressant treatment less than 5 days before inclusion;
* Patient treated in an outpatient setting;
* Patient informed of the diagnosis of his disease;
* Informed patient with written consent.

Exclusion Criteria:

* A current mental or psychiatric impairment or disease (schizophrenia, bipolar disorder) that required psychotropic medication or inpatient treatment on a psychiatric ward;
* A history of psychosis, including schizophrenia, bipolar I or bipolar II disorder, and major depressive disorder with psychotic features;
* Cognitive deficit and not thus being able to comprehend the informed consent and study procedure;
* Patients with somatic, cognitive or other disorders preventing the use of the device (deafness, impaired vision, illiteracy….);
* Non-comprehension of the French language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
A greater clinical response in the active group (smartphone application) comparatively to the comparator group (clinical response was defined as a decline in HDRS-17 score greater than 50%) | Baseline (pre-treatment). 8 weeks post-baseline
  HDRS Hamilton Depressive Rating Scale. Changes in HDRS scores of at least 50% at 8 weeks.

SECONDARY OUTCOMES:
Improvement in scores for therapeutic alliance | baseline (pre-treatment). 8 weeks post-baseline
  Measurement by the 4PAS (4-Point Ordinal Alliance Self-Report)
Improvement in scores for medication adherence | 8 weeks after enrollment
  Measurement by the MARS (Medical Adherence Rating Scale)
Improvement in scores for Quality of Life | 8 weeks after enrollment
  Measurement by the Q-LES-Q-SF (Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Charles PERRENS, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No